CLINICAL TRIAL: NCT05805059
Title: Performance Evaluation of Different Daily Disposable Silicone Hydrogel Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Collaborators: Centre for Ocular Research & Education, Canada (Other)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-145
Record Dates: First submitted 2023-03-28; First posted 2023-04-07 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2023-03

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Contact Lens, Then Test Contact Lens (Experimental): Participants will wear control contact lenses for one week and then crossover to test contact lenses for one week.
  Interventions: Device: Control Contact Lens (stenfilcon A); Device: Test Contact Lens (senofilcon A)
- Test Contact Lens, Then Control Contact Lens (Experimental): Participants will wear test contact lenses for one week and then crossover to control contact lenses for one week.
  Interventions: Device: Control Contact Lens (stenfilcon A); Device: Test Contact Lens (senofilcon A)

INTERVENTIONS:
Device: Control Contact Lens (stenfilcon A) — one week wear
Device: Test Contact Lens (senofilcon A) — one week of wear

SUMMARY:
The goal of this study is to compare the performance of two daily disposable silicone hydrogel contact lenses.

DETAILED DESCRIPTION:
This study is a prospective, bilateral eye, double masked, randomized, 1-week crossover, daily wear design involving two different daily disposable lens types. Each lens type will be worn for approximately one week.

ELIGIBILITY:
Inclusion Criteria:

1. Is between 18 and 35 years of age (inclusively) and has full legal capacity to volunteer;
2. Has read and signed an information consent letter;
3. Self-reports having a full eye examination in the previous two years;
4. Anticipates being able to wear the study lenses for at least 8 hours a day, 7 days a week;
5. Is willing and able to follow instructions and maintain the appointment schedule;
6. Habitually wears soft contact lenses, for the past 3 months minimum;

   1. No more than 1/3 of participants should be habitual wearer of MyDay or MyDay Energys
   2. No more than 1/3 of participants should be habitual wearer of ACUVUE® OASYS MAX 1-Day or ACUVUE® OASYS 1-Day.
7. Has refractive astigmatism no higher than -0.75DC in each eye;
8. Can be fit and achieve binocular distance vision of at least 20/30 Snellen (Available lens parameters are sphere -1.00 to -6.00D, 0.25D steps).

Exclusion Criteria:

1. Is participating in any concurrent clinical or research study;
2. Has any known active ocular disease and/or infection that contraindicates contact lens wear;
3. Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
4. Is using any systemic or topical medications that in the opinion of the investigator may affect contact lens wear or a study outcome variable;
5. Has known sensitivity to the diagnostic sodium fluorescein used in the study;
6. Self-reports as pregnant, lactating or planning a pregnancy at the time of enrolment;
7. Has undergone refractive error surgery or intraocular surgery.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2023-04-14 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sacco, Principal Investigator — Sacco Eye Group, PLLC; Carolyn MacNeil, Principal Investigator — Insight Eye Care; Katherine Bickle, Principal Investigator — ProCare Vision Center; Roxanne Achong-Coan, Principal Investigator — Coan Eye Care
Locations (4):
- United States (3):
  - Coan Eye Care, Ocoee, Florida
  - Sacco Eye Group, PLLC, Vestal, New York
  - ProCare Vision Center, Granville, Ohio
- Insight Eye Care, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Contact Lens, Then Test Contact Lens: Participants wore Control Lens for 1 week (Period 1), and then Test Lens for 1 week (Period 2).
- Test Contact Lens, Then Control Contact Lens: Participants wore Test Lens for 1 week (Period 1), and then Control Lens for 1 week (Period 2).
Period: Period 1 (1 Week)
Arm/Group | Control Contact Lens, Then Test Contact Lens | Test Contact Lens, Then Control Contact Lens
Started | 34 | 34
Completed | 34 | 34
Not Completed | 0 | 0
Period: Period 2 (1 Week)
Arm/Group | Control Contact Lens, Then Test Contact Lens | Test Contact Lens, Then Control Contact Lens
Started | 34 | 34
Completed | 34 | 34
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Analysis Population: All participants who completed study. (Total study population n=68)
Arm/Group | Analysis Population
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27.0 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Lens Handling on Removal
Description: Lens Handling on Removal, using a 0-100 scale (0=Very difficult, 100=Very easy)
Time Frame: Collected once on day 6 at the end of wear
Measure: Mean (Standard Deviation); unit: Units on scale
Groups:
- Control Contact Lens: Participants that received Control Lens during either the first or second period of the study
- Test Contact Lens: Participants that received Test Lens during either the first or second period of the study
Arm/Group | Control Contact Lens | Test Contact Lens
Number analyzed (Participants) | 68 | 68
Units on scale | 95 (12) | 94 (11)

ADVERSE EVENTS:
Time Frame: Duration of the study, approximately 2 weeks.
Description: [Not Specified]
Arm/Group | Control Contact Lens | Test Contact Lens
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/68
Other Adverse Events (participants affected / at risk) | 1/68 | 1/68
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Contact Lens (N=68) | Test Contact Lens (N=68)
eye twitching (Eye disorders) | 1 (1) | 0 (0)
Hyperemia (Eye disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT05805059/Prot_SAP_000.pdf